CLINICAL TRIAL: NCT06960694
Title: Effect of L-carnitine on Disease Activity in Patients With Mild to Moderate Knee Osteoarthritis: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Effect of L-carnitine on Disease Activity in Patients With Mild to Moderate Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Moumita Ghosh, MD Resident (Phase-B), Department of Pharmacology, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMU/2025/5899
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; L-carnitine; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Intervention group) (Experimental)
  Interventions: Drug: L-carnitine
- Group B (Placebo group) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-carnitine — This group will be treated with tablet L-carnitine 330 mg 3 times daily for 8 weeks
  Other Names: Levocarnitine
  Arms: Group A (Intervention group)
Drug: Placebo — This group will be treated with tablet Placebo 330 mg 3 times daily for 8 weeks
  Arms: Group B (Placebo group)

SUMMARY:
The purpose of this study is to evaluate the effects of L-carnitine on symptomatic improvement, oxidative stress, and inflammation in mild to moderate knee osteoarthritis patients.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a progressive degenerative joint disease marked by cartilage degradation, synovial inflammation, and subchondral bone remodeling, resulting in persistent pain and disability. The most prevalent arthritis is OA, and responsible for most adult chronic pain and permanent disability. Osteoarthritis affected 595 million individuals worldwide in 2020, which accounted for 7.6% of the world's population. The most common kind of OA is knee osteoarthritis. Currently, there is no safe and effective therapy for knee OA. Nonsteroidal anti-inflammatory medicines are commonly used to treat the symptoms of osteoarthritis, but long-term usage can lead to renal and cardiac complications. There is a higher demand for medicine that not only relieve symptoms but also decrease disease progression. Recently, there has been an increase in interest in complementary and alternative therapies, particularly nutritional supplements. L-carnitine, a naturally occurring chemical, is required for carrying long-chain fatty acids to the mitochondria, where they are oxidized to generate energy. It is mostly generated in the liver and kidneys from the amino acids-lysine and methionine. Research has demonstrated that L-carnitine has anti-inflammatory and antioxidant characteristics. Several animal and human studies have indicated that it improves osteoarthritis by lowering oxidative stress and inflammation. The proposed study aims to determine whether L-carnitine is more effective in lowering disease activity in mild to moderate knee OA compared to placebo. It will be a single-center study, utilizing a double-blind, randomized placebo-controlled trial design. The study will involve 66 patients with mild to moderate knee OA. The participants will be randomly be assigned into two groups: Intervention group and Placebo group. Patients of Intervention group will receive tablet L-carnitine 330 mg 3 times daily for 8 weeks. The patients of Placebo group will receive tablet placebo 330 mg 3 times daily for the 8 weeks. In this study, we will evaluate MDA (Malondialdehyde), GSH (Glutathione), and hs-CRP (high-sensitivity C-reactive protein) concentrations and three dimensions (pain, stiffness and physical activity) of Bangla version of WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index). In addition, we will assess various sociodemographic characteristics of all the participants.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain
* Radiographic evidence of mild to moderate knee osteoarthritis (Kellgren-Lawrence Grade: II-III)
* Above 40 years
* Both male and female

Exclusion Criteria:

* Chronic kidney disease or chronic liver disease
* Diagnosed with systemic inflammatory disorders, such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, gout
* Patients on immunosuppressant treatment
* Any history of intra-articular corticosteroid injections during the previous 2 months
* A history of knee surgery or trauma
* Any antioxidant vitamins use, such as A, C, and E, or history of use in the last two months
* History of taking L-carnitine and NSAIDs in last 2 months
* Pregnancy or lactation
* Participation in another clinical trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2025-06-28 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
Pain, stiffness and physical function | 8 weeks
  To assess and compare pain, stiffness and physical function in mild to moderate knee osteoarthritis patients, a translated and validated Bangla version of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) VA3.01 will be used

SECONDARY OUTCOMES:
Oxidative stress markers (Malondialdehyde and Glutathione) | 8 weeks
Inflammatory marker (hs-CRP) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Moumita Ghosh, MBBS, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided